CLINICAL TRIAL: NCT04090281
Title: Implementing Precision Medicine Approaches to Guide Anti-platelet Selection Following Percutaneous Coronary Intervention (PCI)
Brief Title: Implementing Precision Medicine Approaches to Guide Anti-platelet Selection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Scott Mosley, PharmD, Assistant Professor of Clinical Pharmacy, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-19-00099
Record Dates: First submitted 2019-09-06; First posted 2019-09-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Acute Coronary Syndrome (ACS); STEMI - ST Elevation Myocardial Infarction (MI); NSTEMI - Non-ST Segment Elevation MI; Unstable Angina (UA)
Keywords: precision medicine; antiplatelet; pharmacogenetics; de-escalation; dual antiplatelet therapy (DAPT); percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single arm, pragmatic study to determine feasibility of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Precision medicine implementation (Other): Patients will receive a precision medicine approach, incorporating both CYP2C19 genotyping and platelet reactivity phenotyping, to guide dual antiplatelet therapy selection for patients with ACS, post PCI and followed over a 12 month period.
  Interventions: Genetic: CYP2C19 genotyping

INTERVENTIONS:
Genetic: CYP2C19 genotyping — Upon hospital discharge, patients will undergo CYP2C19 genotyping to guide initial P2Y12 inhibitor selection. At 14 days, post discharge, patients will undergo on treatment platelet reactivity phenotyping to further guide deescalation of P2Y12 inhibitor therapy
  Other Names: platelet reactivity phenotyping

SUMMARY:
The study aims to determine the feasibility and clinical utility of incorporating precision medicine approaches, incorporating both cytochrome P450 2C19 (CYP2C19) genotyping and platelet reactivity phenotyping, with standard of care for patients with acute coronary syndromes (ACS), post PCI.

DETAILED DESCRIPTION:
Study Population:

Adult patients will be eligible for inclusion if they provide informed consent and have no contraindications for 12-months of dual antiplatelet therapy (DAPT).

Baseline Evaluation:

Overview of clinical protocol: Patients with successful PCI will receive a genotype guided recommendation, upon discharge, based on CYP2C19 genotype. Patients who are determined to have CYP2C19 poor metabolizer (PM) or intermediate metabolizer (IM) status will be recommended to receive 12-months of prasugrel. Patients who are determined to have CYP2C19 normal metabolizer (NM), rapid metabolizer (RM), or ultra-rapid metabolizer (UM) phenotype will be recommended to receive a de-escalation treatment, guided by on-treatment platelet reactivity phenotype at 14 days, post discharge.

30-day, 6-month, and 12-month Follow-up: Patients will be contacted by phone or visited during one of their regularly scheduled appointments, at 14 days, 30 days, 6 months , and 12 months, to complete "Follow-up Case Report Forms" to collect outcomes data. The 12-month follow up communication with enrolled patients will end their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with troponin positive ACS
2. Patients scheduled for left heart catheterization and undergoing PCI
3. Age 18-80 years at time of enrollment
4. Currently receiving or anticipated to receive DAPT, with P2Y12 inhibitor
5. Ability to follow-up for a clinic visit with LAC+USC outpatient cardiology
6. Written informed consent

Exclusion Criteria:

1. Subjects with known contraindications to clopidogrel treatment, which are hypersensitivity to the drug substance or any component of the product and active pathological bleeding such as peptic ulcer or intracranial hemorrhage
2. Subjects with known contraindications to prasugrel treatment, which are hypersensitivity to the drug substance or any component of the product, active pathological bleeding such as peptic ulcer or intracranial hemorrhage, and a history of prior transient ischemic attack (TIA) or stroke
3. Subjects with a history of a complicated or prolonged cardiogenic shock in the last two weeks prior to enrolling in this study. A complicated or prolonged cardiogenic shock is defined by a cardiogenic shock that required mechanical ventilation or the cardiovascular support with positive inotropic drugs (i. v. catecholamines) for ≥7 days.
4. Subjects requiring concomitant treatment with an anticoagulant agent (Vitamin-K antagonists or novel oral anticoagulants such as rivaroxaban, dabigatran or apixaban)
5. Indication for major surgery (per decision of the treating physician) for the planned duration of the study
6. Subject with history of liver transplant or plan to undergo liver transplant during the next 12 months
7. Evidence of significant active neuropsychiatric disease, in the investigator's opinion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing pharmacogenetics to guide antiplatelet therapy | 12 months
  The proportion of patients in whom a genetic-guided recommendation is accepted by the clinician
Feasibility of implementing platelet reactivity testing to guide de-escalation of antiplatelet therapy | 12 months
  The proportion of patients in whom a platelet reactivity phenotype-guided recommendation is accepted by the clinician

SECONDARY OUTCOMES:
Net clinical utility | 30 days
  The incidence of combined endpoints of major adverse cardiovascular events (MACE), stent thrombosis, unstable angina, major and minor bleeding, all-cause mortality, and hospital readmission rate within 30 days, post discharge
Net clinical utility | 12 months
  The incidence of combined endpoints of MACE, stent thrombosis, unstable angina, major and minor bleeding, all-cause mortality, and hospital readmission rate within 12 months, post discharge
Change in score of anxiety using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 30 days
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for anxiety include fear, anxiety, worry, and uneasiness. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.
Change in score of anxiety using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for anxiety include fear, anxiety, worry, and uneasiness. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.
Change in score of depression using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 30 days
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for depression include worthless, helpless, depressed, and hopelessness. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.
Change in score of depression using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for depression include worthless, helpless, depressed, and hopelessness. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.
Change in score of social abilities using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 30 days
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for social abilities include leisure, family, usual work, and friends. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.
Change in score of social abilities using (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for social abilities include leisure, family, usual work, and friends. A score of 0 to 20 based on survey responses will be resulted for this subscale, with higher values representing a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Mosley, PharmD, Principal Investigator — University of Southern California School of Pharmacy
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Study protocol is anticipated to be published within 12 months of completing the study, and not anticipated to have a time limit.